CLINICAL TRIAL: NCT05274906
Title: Red and Processed Meat Effects on the Metabolome and Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Marian Neuhouser, Faculty Member, Program Head, Cancer Prevention Program, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: RG1121543; 1R21DK128754-01 (NIH)
Record Dates: First submitted 2022-02-18; First posted 2022-03-11 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Controlled Feeding Trial; Healthy Eating Index; Red Meat; Meat
MeSH Terms: interventions — Random Allocation; Diet; Dyrk Kinases; Methods

STUDY DESIGN:
Intervention Model Description: Randomized cross-over
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controlled HEI-2015-M diet, followed by controlled HEI-2015 diet. (Experimental): Participants first complete a 21-day controlled HEI-2015 diet with red and processed meat (HEI-2015-M). After a washout period of 1 week or longer, participants then complete the same 21-day controlled HEI-2015 diet without red and processed meat (HEI-2015)
  Interventions: Other: Randomized, cross-over controlled feeding trial testing a Healthy Eating Index 2015 (HEI-2015) diet with and without red and processed meat
- Controlled HEI-2015 diet, followed by controlled HEI-2015-M diet. (Experimental): Participants first complete a 21-day controlled HEI-2015 diet without red and processed meat (HEI-2015). After a washout period of 1 week or longer, participants then complete the same 21-day controlled HEI-2015 diet with red and processed meat (HEI-2015-M).
  Interventions: Other: Randomized, cross-over controlled feeding trial testing a Healthy Eating Index 2015 (HEI-2015) diet with and without red and processed meat

INTERVENTIONS:
Other: Randomized, cross-over controlled feeding trial testing a Healthy Eating Index 2015 (HEI-2015) diet with and without red and processed meat — Healthy Eating Index-2015 (HEI-2015) with or without red/processed meat (HEI-2015-M)
  Other Names: feeding trial, intervention, dietary, HEI-2015

SUMMARY:
This controlled feeding trial will identify biomarkers in the metabolome and microbiome that may differ when consuming a healthy diet with or without red and processed meat.

DETAILED DESCRIPTION:
This is a randomized cross-over feeding trial to test whether red and processed meat consumption, in the context of a controlled diet based on HEI-2015, will cause shifts in the metabolome and the microbiome compared to a controlled HEI-2015 diet with no red or processed meat. Twenty healthy adult volunteers will consume two diets in random order: 1) Diet A is based on the Healthy Eating Index-2015 (HEI-2015) and includes no red or processed meat; 2) Diet B is based on the Healthy Eating Index-2015 and includes red and processed meat (HEI-2015-M) as some of the protein sources. Both diet periods last 21 days and an approximately 21-day washout period occurs between diets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult,
* 18-50 years of age,
* able to read, speak, and understand English, and
* willing to come to the Fred Hutchinson Cancer Research Center campus twice weekly during study

Exclusion Criteria:

* known allergy to red or processed meat,
* vegetarian or vegan,
* any religious or personal reason(s) to avoid red and processed meat,
* pregnant an/or exclusively breastfeeding, and/or
* alcohol or recreational drug abuse

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marian L. Neuhouser, PhD, RD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Controlled HEI-2015 Diet, Followed by Contrilled HEI-2015-M Diet.: Participants first complete a 21-day controlled HEI-2015 diet without red and processed meat (HEI-2015). After a washout period of 1 week or longer, participants then complete the same 21-day controlled HEI-2015 diet with red and processed meat (HEI-2015-M).
Period: Overall Study
Arm/Group | Controlled HEI-2015-M Diet, Followed by Controlled HEI-2015 Diet. | Controlled HEI-2015 Diet, Followed by Contrilled HEI-2015-M Diet.
Started | 12 | 11
Completed | 10 | 10
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: Age in years at time of enrollment based on participant-reported questionnaire
Groups:
- Total: Total of all reporting groups
Arm/Group | Controlled HEI-2015-M Diet, Followed by Controlled HEI-2015 Diet. | Controlled HEI-2015 Diet, Followed by Contrilled HEI-2015-M Diet. | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 34 [26 to 49] | 34 [22 to 50] | 34 [22 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 10 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Test the Effects of Red and Processed Meat on Aqueous Biomarkers of the Blood Metabolome
Description: Plasma aqueous metabolomics were evaluated via Liquid Chromatography/Mass Spectrometry (LC/MS). Data are relative concentrations - the concentration of a specified biomarker is relative to the concentration of all other biomarkers. Data are reported as the mean ratio of relative concentration on day 21 compared to day 0 [(relative concentration day 21)/(relative concentration day 0)]. A value above 1.0 indicates that the relative concentration of the metabolite increased from baseline at the end of the diet, whereas a value below 1.0 indicates the relative concentration decreased, and a value of 1.0 indicates no change from baseline.
Time Frame: Day 21
Population: Cross-over design; each participant completed each arm in random order
Measure: Mean (Standard Deviation); unit: ratio of day 21 to day 0
Groups:
- Controlled HEI-2015-M: Controlled HEI-2015 diet with red and processed meat.
- Controlled HEI-2015: Controlled HEI-2015 diet without red and processed meat
Arm/Group | Controlled HEI-2015-M | Controlled HEI-2015
Number analyzed (Participants) | 20 | 20
ratio of day 21 to day 0
  Hydroxyproline | 0.87 (0.43) | 0.60 (0.30)
  1/3-Methylhistidine | 3.48 (4.50) | 5.66 (7.55)
  Acetylcarnitine | 0.99 (0.24) | 0.88 (0.24)
  Lactose/Trehalose | 1.17 (0.61) | 0.91 (0.49)
  N-AcetylGlycine | 1.36 (0.98) | 1.10 (0.62)
  Cis-Aconitate | 1.05 (0.33) | 0.89 (0.34)

2. Primary Outcome: Test the Effects of Red and Processed Meat on Lipid Biomarkers of the Blood Metabolome
Description: Plasma lipid metabolomics were evaluated via Liquid Chromatography/Mass Spectrometry (LC/MS). Data are absolute concentrations. Data are reported as the mean ratio of relative concentration on day 21 compared to day 0 [(relative concentration day 21)/(relative concentration day 0)]. A value above 1.0 indicates that the relative concentration of the metabolite increased from baseline at the end of the diet, whereas a value below 1.0 indicates the relative concentration decreased, and a value of 1.0 indicates no change from baseline.
Time Frame: Day 21
Population: Cross-over design; each participant completed each arm in random order
Measure: Mean (Standard Deviation); unit: ratio of day 21 to day 0
Arm/Group | Controlled HEI-2015-M | Controlled HEI-2015
Number analyzed (Participants) | 20 | 20
ratio of day 21 to day 0
  Cholesterol Esther 20:5 | 1.09 (0.67) | 0.98 (0.58)
  Lysophosphatidylethanolamine 20:3 | 1.11 (0.34) | 0.97 (0.29)
  Lysophosphatidylethanolamine 22:5 | 0.89 (0.29) | 0.80 (0.18)
  Phosphatidylcholine 18:0/20:5 | 1.11 (1.14) | 0.90 (0.83)
  Phosphatidylethanolamine P-18:0/20:3 | 1.10 (0.47) | 0.88 (0.33)
  Phosphatidylethanolamine P-18:1/18:2 | 0.82 (0.24) | 0.65 (0.20)
  Phosphatidylethanolamine P-18:0/20:5 | 0.80 (0.48) | 0.59 (0.28)
  Triacylglycerol 51:2-FA16:0 | 1.42 (1.56) | 1.39 (1.86)
  Triacylglycerol 54:7-FA22:5 | 1.37 (0.75) | 1.62 (0.88)
  Cholesterol Esther 18:3 | 1.00 (0.31) | 0.90 (0.28)
  Ceramides d18:1(24:0) | 0.90 (0.18) | 0.84 (0.20)
  Diacylglycerol 18:2/20:4 | 1.15 (0.19) | 1.31 (0.66)
  Hexosylceramides d18:1(22:0) | 0.88 (0.14) | 0.82 (0.13)
  Lysophosphatidylcholine (19:0) | 1.13 (0.30) | 1.05 (0.31)
  Lysophosphatidylethanolamine 20:2 | 0.79 (0.22) | 0.68 (0.19)
  Phosphatidylcholine 16:0/20:5 | 1.06 (0.83) | 0.89 (0.57)
  Phosphatidylcholine 18:0/20:3 | 1.12 (0.41) | 1.01 (0.39)
  Phosphatidylcholine 18:2/20:3 | 1.10 (0.33) | 0.94 (0.29)
  Phosphatidylethanolamine O-16:0/22:6 | 1.13 (0.51) | 0.94 (0.37)
  Phosphatidylethanolamine P-16:0/18:1 | 0.93 (0.28) | 0.83 (0.21)
  Phosphatidylethanolamine P-16:0/18:2 | 0.88 (0.31) | 0.77 (0.23)
  Phosphatidylethanolamine P-16:0/22:5 | 0.90 (0.25) | 0.79 (0.21)
  Phosphatidylethanolamine P-18:0/18:1 | 0.84 (0.23) | 0.72 (0.17)
  Phosphatidylethanolamine P-18:0/18:2 | 0.82 (0.27) | 0.67 (0.19)
  Phosphatidylethanolamine P-18:0/20:4 | 1.10 (0.44) | 0.97 (0.37)
  Phosphatidylethanolamine P-18:0/22:5 | 0.89 (0.28) | 0.78 (0.29)
  Phosphatidylethanolamine P-18:1/18:1 | 0.84 (0.27) | 0.68 (0.20)
  Phosphatidylethanolamine P-18:1/20:4 | 1.11 (0.44) | 0.95 (0.35)
  Phosphoinositides 18:0/18:1 | 0.93 (0.37) | 0.82 (0.30)
  Triacylglycerol 54:8-FA22:6 | 1.36 (0.74) | 1.78 (1.14)

3. Primary Outcome: Test the Effects of Red and Processed Meat on Biomarkers on the Urine Metabolome
Description: Effects of the intervention on urine metabolomic biomarkers were evaluated via Nuclear Magnetic Resonance (NMR). Urine metabolites are absolute concentrations standardized (as a ratio) to trimethyl-silylpropionic-2,2,3,3-d4 acid sodium salt (TSP). Data are reported as the mean ratio of relative concentration on day 21 compared to day 0 [(relative concentration day 21)/(relative concentration day 0)]. A value above 1.0 indicates that the relative concentration of the metabolite increased from baseline at the end of the diet, whereas a value below 1.0 indicates the relative concentration decreased, and a value of 1.0 indicates no change from baseline.
Time Frame: Day 21
Population: Cross-over design; each participant completed each arm in random order
Measure: Mean (Standard Deviation); unit: ratio of day 21 to day 0
Arm/Group | Controlled HEI-2015-M | Controlled HEI-2015
Number analyzed (Participants) | 20 | 20
ratio of day 21 to day 0
  Citrate | 0.99 (0.61) | 1.09 (0.42)
  Allantoin | 1.54 (0.96) | 2.18 (1.41)
  3_hydroxyisovaleric acid | 1.16 (0.70) | 1.24 (0.41)
  Glucose | 1.10 (0.63) | 1.22 (0.45)
  Creatine | 1.21 (0.80) | 0.90 (0.42)
  2_Oxoglutarate | 1.17 (1.31) | 1.11 (0.36)
  Choline | 1.34 (1.01) | 1.12 (1.59)
  Ascorbic Acid | 2.59 (3.16) | 3.02 (3.53)
  Propanediol | 2.60 (4.62) | 3.43 (4.91)

4. Primary Outcome: Test the Effects of Red and Processed Meat on Gut Microbiome
Description: Shannon's Diversity Index (SDI) was used as a measure of species diversity, calculated as the sum of -p/ln(p), where p is the proportion of the sample made up of each OTU using the QIIME2 shannon_pd plugin. Sampled 16S rRNA sequences were organized into 'amplicon sequence variants' (ASVs), ASVs were filtered by abundance with a threshold of 1e - 5. This measure is a unitless scale proportion ranging from zero to infinity. Zero indicates a completely homogenous sample, and higher scores indicate greater species diversity.
Time Frame: Day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Controlled HEI-2015-M | Controlled HEI-2015
Number analyzed (Participants) | 20 | 20
score on a scale | 0.99 (0.10) | 1.00 (0.07)

5. Primary Outcome: Test the Effects of Red and Processed Meat on Fecal Bacterial Functional Genes
Description: Fecal bacterial functional genes were evaluated via digital droplet PCR. Data are reported as the difference between day 21 and day 0 (calculated as day 21 - day 0) of each diet in the relative abundance (calculated as gene counts/16s rRNA gene counts) of fecal bacterial functional genes. A value that is positive indicates that the relative abundance increased from baseline to the end of the diet, whereas a negative value indicates the relative abundance decreased.
Time Frame: Day 21
Measure: Mean (Standard Deviation); unit: proportion of gene counts
Arm/Group | Controlled HEI-2015-M | Controlled HEI-2015
Number analyzed (Participants) | 20 | 20
proportion of gene counts
  Butyryl-CoA:acetate CoA transferase (in bacteria species Roseburia) | 0.54 (1.9) | 0.24 (1.3)
  Butyryl-CoA:acetate CoA transferase (in bacteria species Eubacteirum rectale) | 0.07 (0.4) | 0.19 (0.6)
  Nitrate reductase (in bacteria species Escherichia/Shigella) | 0.23 (0.5) | 0.11 (0.3)

ADVERSE EVENTS:
Time Frame: From start of intervention to ending of intervention: up to 9 weeks
Description: Method of assessment: participant reported via interview with study staff at each clinic visit
Groups:
- Controlled HEI-2015-M Diet: 21-day controlled HEI-2015 diet with red and processed meat (HEI-2015-M).
- Controlled HEI-2015 Diet: 21-day controlled HEI-2015 diet without red and processed meat (HEI-2015).
Arm/Group | Controlled HEI-2015-M Diet | Controlled HEI-2015 Diet
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/06/NCT05274906/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT05274906/ICF_001.pdf